CLINICAL TRIAL: NCT06029582
Title: The Use of Virtual Reality Headset in Controlling Pain During Pregnancy Termination; a Randomized Control Trial
Brief Title: VR Headset for Pain During Pregnancy Termination
Acronym: VRPASAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLIR-2023-55
Record Dates: First submitted 2023-06-20; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy Termination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality headset (Experimental): Individuals will wear the Virtual Reality Headset that produce a calming scenario
  Interventions: Device: VR headset
- controls (No Intervention): no headset

INTERVENTIONS:
Device: VR headset — Virtual Reality Headset
  Arms: Virtual Reality headset

SUMMARY:
The goal of this randomized control study is to see if virtual reality headsets (VRHS) are useful in women undergoing surgical pregnancy termination. The main questions it aims to answer are:

Do VRHS decrease the pain associated with surgical pregnancy termination Participants will wear the VRHS during the surgery and take a pain survey before and after the procedure. The pain assessment will be compared to placebo headset which will be randomly assigned.

DETAILED DESCRIPTION:
Use of virtual reality headsets have been employed in cancer and behavioral medicine fields with moderate success in controlling anxiety stress and pain. The decision to terminate a pregnancy can create significant stress and anxiety. In the US, there are over 900,000 pregnancy terminations each year with many patients undergoing dilation and evacuation with minimal anesthesia. We plan to assess virtual reality headset's ability to decrease pain associated with surgical termination of pregnancy.

Patient's will be recruited from a single outpatient family-planning center. Inclusion criteria include all patients over the age of 18 that are undergoing a surgical termination of pregnancy in the first and second trimester under local and/or conscious sedation anesthesia. Patients under the age of 18 with significant medical comorbidities will be excluded. Patient demographics including age, BMI, obstetric/ gynecology history, and prior terminations will be collected. Patients will be given pre- procedure survey to assess anxiety and stress. The survey will be self-administered with assistance from study personnel. Patients will then be randomized to either the virtual reality headset or no headset. The procedure will be then performed with the headsets on the patients. Amount and type of local anesthesia employed will be recorded. After the procedure (within 1 hour), the individuals will be resurveyed for both stress and anxiety, with the addition of a visual analog scale to assessing pain associated with the procedure. Pre and post vital signs will also be extracted from the chart. The patient as well as the clinician performing the procedure will be masked as to the intervention. We will require 50 patients per arm assuming a 30% reduction in the pain scale (power 80%, 95% CI, with SD of 0.70). Logistic regression will be performed for those comorbidities that may be influence our outcome, such as age, BMI, prior terminations.

ELIGIBILITY:
Inclusion Criteria:

* all healthy patients undergoing a first or second trimester pregnancy termination

Exclusion Criteria:

* pregnancy patients requesting a termination under the age of 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-08 (Estimated); Study Completion 2024-07-07 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | immediately after procedure (10 minutes)
  A pain scale (visual analog scale) will be used to assess reduction of pain (scale 1-10) one being no pain, 10 highest level of pain

SECONDARY OUTCOMES:
Anxiety reduction | pre and post procedure 1 hr before procedure and within 10 minutes after
  A scale will be used to assess anxiety (Visual analog scale: scale 1-10) 1 being no stress, 10 being highest level of stress

OTHER OUTCOMES:
Heart rate variation | pre and post procedure, 10 minutes before and 10, 20 minutes after
  Changes in heart rate in beats per minute
Blood pressure variation | pre and post procedure, 10 minutes before and 10, 20 minutes after
  Changes in blood Pressure (mm/Hg)

CONTACTS AND LOCATIONS:
Overall Officials: James N Anasti, MD, Principal Investigator — St Luke's University Hosptial
Locations (1):
- Allentown Women Center, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No